CLINICAL TRIAL: NCT03532841
Title: Role of Oral Tramadol 50 mg in Reducing Pain During Colposcopy-directed Cervical Biopsy: A Randomised Double-blind Placebo-controlled Trial
Brief Title: Role of Oral Tramadol 50 mg in Reducing Pain During Colposcopy-directed Cervical Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology,faculty of medicine,Cairo university., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: tramadol and colposcopy
Record Dates: First submitted 2018-04-13; First posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Cervical Biopsy
MeSH Terms: interventions — Tramadol; Tablets

STUDY DESIGN:
Intervention Model Description: A randomised double-blind placebo-controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (tramadol group) (Experimental): Group I will receive an oral tramadol 50 mg(Tramal, Memphis, Giza, Egypt) tablet one hour before the procedure.
  Interventions: Drug: an oral tramadol 50 mg(Tramal, Memphis, Giza, Egypt) tablet
- Group II (placebo oral tablet group) (Placebo Comparator): group II will receive a placebo one hour before the procedure.the Treatment and placebo will be identical in form and packaging, without any identifying label.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: an oral tramadol 50 mg(Tramal, Memphis, Giza, Egypt) tablet — Group I will receive an oral tramadol 50 mg(Tramal, Memphis, Giza, Egypt) tablet one hour before the procedure.
  Arms: Group I (tramadol group)
Drug: Placebo Oral Tablet — placebo tablet of the same shape,color and taste will be given in the placebo arm
  Other Names: placebo comparator or group II
  Arms: Group II (placebo oral tablet group)

SUMMARY:
The study objective is to evaluate the effectiveness of oral tramadol 50 mg in reducing pain during the colposcopy-directed cervical biopsy.half of the patients will receive oral tramadol tablets and the other half will receive a placebo.

DETAILED DESCRIPTION:
.Colposcopy-directed cervical biopsy (CDB) is a procedure performed in women with abnormal Papanicolaou smear or abnormal human papillomavirus (HPV) testing whose cervical lesions are colposcopically identified. Generally, no anaesthesia is needed for the procedure which can be done on an outpatient basis.The degree of pain associated with this procedure varies from mild to severe and many studies suggested that pain levels are often high reaching a score of more than 40 points on a 100-point visual analogue scale (VAS). Tramadol hydrochloride is an orally active centrally acting synthetic opioid. It is an atypical analgesic with a dual mechanism of action: serotonin and norepinephrine reuptake inhibition and modest l-opioid agonist. It has a lower incidence of respiratory depression, cardiac depression, side effects on smooth muscle and abuse potential as compared to typical opioid agents

ELIGIBILITY:
Inclusion Criteria:

Women with abnormal cervical cytology candidate for colposcopy and colposcopically directed biopsy or loop electrosurgical excision procedure.

Exclusion Criteria:

* Patients taking psychotropic or anticoagulant medications or with histories of bleeding disorders or bleeding ulcers.
* Cervical and vaginal infection
* pregnant patients.
* Patients who had taken analgesics in the previous 24 hours, had a history of drug abuse or allergy to tramadol or opioids
* Patients with contraindications to tramadol as severe asthma, severe renal or hepatic impairment, People with uncontrolled epilepsy.
* People under the influence of (intoxicated with) alcohol, sleeping tablets, tranquilisers, psychotropic drugs (those affecting mood or emotions) or other opioid painkillers, e.g. morphine, codeine.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2018-05-15 (Estimated); Primary Completion 2018-08-20 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
patient-described pain level | immediately after speculum placement (baseline pain score).
  the mean patient-described pain level will be measured with the visual analogue scale (VAS). Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10. A higher score indicates greater pain intensity. Subjects will be told that the far left point will represent "no pain "and the far right point will represent "the worst pain you can imagine." They will be asked to mark a vertical line on the visual analogue scale during the procedure to note levels of discomfort.
patient-described pain level | after the ﬁrst ectocervical biopsy(approximately 5 minutes after speculum insertion)
  the visual analogue scale score from 0-10
patient-described pain level | the overall pain at 30 min after the procedure (postprocedure pain score)
  (postprocedure pain score) using the visual analogue scale score from 0-10.

SECONDARY OUTCOMES:
duration of colposcopy procedure. | from speculum insertion to colposcopy removal at the end of procedure.
  relationship between pain score and colposcopy duration in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided